CLINICAL TRIAL: NCT07281768
Title: Combining Capecitabine/Oxaliplatin Chemotherapy With Cemiplimab Alone or in Combination With Fianlimab or REGN7075 for the Neoadjuvant Treatment of Locally Advanced Rectal Cancer
Brief Title: Capecitabine/Oxaliplatin Chemotherapy and Cemiplimab With or Without Fianlimab or REGN7075 in Locally Advanced Rectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J25118; IRB00505702 (Other: Johns Hopkins Medical Institution)
Record Dates: First submitted 2025-12-04; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
Keywords: Rectal Cancer; Cemiplimab; Fianlimab; REGEN7075; Oxaliplatin; Capecitabine; Immunotherapy; Anti-PD-1 (Programmed Death-Ligand 1)(protein immune checkpoint); PD-L1 (Programmed Death-Ligand 1)(protein immune checkpoint); Adenocarcinoma; Carcinoma; CAPOX; Chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms; Adenocarcinoma; Carcinoma | interventions — Oxaliplatin; Capecitabine; cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Oxaliplatin, Capecitabine, Cemiplimab) (Experimental)
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Cemiplimab
- Arm B (Oxaliplatin, Capecitabine, Cemiplimab, Fianlimab) (Experimental)
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Cemiplimab; Drug: Fianlimab
- Arm C (Oxaliplatin, Capecitabine, Cemiplimab, REGN7075) (Experimental)
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Cemiplimab; Drug: REGN7075

INTERVENTIONS:
Drug: Oxaliplatin — Patients will receive Oxaliplatin (130mg/m^2 administered IV) on Day 1 of each 21 day cycle for a total of 4 cycles of treatment.
Drug: Capecitabine — Patients will receive Capecitabine (1000mg/m^2 administered orally) on Days 1 through 14 of each 21 day cycle for a total of 4 cycles of treatment.
  Other Names: Xeloda
Drug: Cemiplimab — Patients will receive Cemiplimab (350 mg administered IV) on Day 1 of each 21 day cycle for a total of 4 cycles of treatment.
  Other Names: REGN2810; LIBTAYO
Drug: Fianlimab — Patients will receive Fianlimab (1600 mg administered IV) on Day 1 of each 21 day cycle for a total of 4 cycles of treatment.
  Other Names: REGN3767
  Arms: Arm B (Oxaliplatin, Capecitabine, Cemiplimab, Fianlimab)
Drug: REGN7075 — Patients will receive REGN7075 (2700 mg administered IV) on Day 1 of each 21 day cycle for a total of 4 cycles of treatment.
  Arms: Arm C (Oxaliplatin, Capecitabine, Cemiplimab, REGN7075)

SUMMARY:
The purpose of this study is to evaluate the safety and clinical activity of combining cemiplimab, cemiplimab/fianlimab, or cemiplimab/REGN7075 with capecitabine/oxaliplatin (CAPOX) for the neoadjuvant treatment of patients with microsatellite stable (MSS) locally advanced rectal cancer (T2 node-positive, T3 node-negative, T3 node-positive).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1.
* Rectal cancer (with tumor tissue present at or below the peritoneal reflection) as determined by MRI pelvis or endoscopic ultrasound.
* Have histologically proven mismatch repair proficient (pMMR) or microsatellite stable (MSS) rectal adenocarcinoma.
* Must not have received any prior systemic treatment or radiation.
* Candidate for sphincter-sparing surgical resection after neoadjuvant therapy according to the primary surgeon.
* Patients have the following clinical staging:

  * cT2 node-positive:
  * T: Tumor is invading the muscularis propria but has not grown through it to the serosa
  * N: At least 1 perirectal lymph node ≥5 mm and no more than 4 perirectal lymph nodes >10 mm in short axis
  * M: No evidence of metastasis
  * cT3 node-negative
  * T: Tumor has grown through the muscularis propria into the serosa but has not invaded nearby organs
  * N: No perirectal lymph nodes ≥ 5 mm in size that suggest tumor involvement
  * M: No evidence of metastasis
  * cT3 node-positive
  * T: Tumor has grown through the muscularis propria into the serosa but has not invaded nearby organs
  * N: At least 1 perirectal lymph node ≥ 5 mm and no more than 4 perirectal lymph nodes > 10 mm in size in short axis
  * M: No evidence of metastasis
* Absence of distant metastases on CT or MRI imaging
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests and procedures.
* LVEF assessment with documented LVEF ≥ 50% by either TTE or MUGA (TTE preferred) within 6 months from first study drug administration.
* For both Women and Men, must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Have received an investigational agent or used an investigational device within 28 days of the first dose of study drug.
* Have expected to require any other form of systemic or localized antineoplastic therapy while on study.
* Have had surgery within 28 days of dosing of investigational agent, excluding minor procedures (dental work, skin biopsy, etc.).
* History of prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA4, or anti-Lag-3 antibodies for any reason.
* Currently using any chronic systemic steroids.
* History of severe hypersensitivity reaction to any monoclonal antibody.
* History of encephalitis, meningitis, dementia, Parkinson's or uncontrolled seizures within 1 year prior to the first dose of study drug.
* Uncontrolled infection of HIV, HBV, HCV, or Tuberculosis.
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, metastatic cancer, or psychiatric illness/social situations that would limit compliance with study requirements.
* Active autoimmune disease.
* Any tissue or organ allograft, regardless of need for immunosuppression, including corneal allograft.
* Patient has a pulse oximetry of <92% on room air.
* Patient is on supplemental home oxygen.
* Has clinically significant heart disease.
* Troponin T (TnT) or troponin I (TnI) > 2x institutional ULN at baseline.
* Conditions, including alcohol or drug dependence, intercurrent illness, or lack of sufficient peripheral venous access, that would affect the patient's ability to comply with study visits and procedures.
* Patient is pregnant or breastfeeding.
* Unwilling or unable to follow the study schedule for any reason.
* Patient received a live vaccine within 30 days of planned start of study medication.
* Receipt of COVID-19 vaccination within 1 week of planned start of study medication or for which the planned COVID-19 vaccinations would not be completed 1 week prior to start of study medication.
* Patients with T4 disease or N2 disease (as defined by >/= 4 lymph nodes, each greater or equal to 10 mm in short axis).
* Evidence that the tumor is adjacent to (defined as within 3 mm of) the mesorectal fascia on pre-operative MRI or endorectal ultrasound or pelvic CT scan.
* Patients with symptomatic untreated bowel obstruction due to rectal cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) rate | 24 months
  Proportion of subjects with a pathologic complete response (pCR) at the time of surgery. pCR is defined as subjects with no viable tumor cell noted on pathological evaluation of the resection specimen using the College of American Pathologists (CAP) tumor regression scoring system (CAP tumor regression score of 0).

SECONDARY OUTCOMES:
Number of participants experiencing grade 3 or above drug-related toxicities | 12 weeks
  When calculating the incidence of Adverse Events (AEs), each AE (as defined by NCI CTCAE v6.0) will be counted only once for a given subject.
Pathologic Response Rate | 24 months
  Pathologic response rate as defined as the proportion of subjects with complete or partial tumor regression at the time of surgery using the College of American Pathologists (CAP) tumor regression scoring system (CAP tumor regression score of 0 to 2).
Event-free Survival (EFS) | 24 months
  EFS is defined as the number of months from the date of initiation of neoadjuvant treatment to disease relapse or development of metastatic disease (as assessed using RECIST 1.1 criteria) or death due to any cause. EFS will be censored at the date of the last scan for subjects without documentation of disease progression at the time of analysis.
Composite Complete Response Rate | 24 months
  Composite complete response rate is defined as the proportion of subjects with either a pathologic complete response (pCR) or those that remain disease-free for 24 months on radiographic imaging and endoscopic evaluation for those that elected to not go to surgery. pCR is defined as subjects with no viable tumor cell noted on pathological evaluation of the resection specimen using the College of American Pathologists (CAP) tumor regression scoring system (CAP tumor regression score of 0).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Christenson, MD, Principal Investigator — Johns Hopkins Sidney Kimmel Comprehensive Cancer Center
Locations (1):
- Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No